CLINICAL TRIAL: NCT02255448
Title: Evaluation of the esCCO Non-invasive Cardiac Output Measurement Device in Pregnancy
Acronym: esCCO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single
Other Study IDs: 14/YH/1182
Record Dates: First submitted 2014-09-30; First posted 2014-10-02 (Estimated); Last update posted 2014-10-03 (Estimated); Status verified 2014-09

CONDITIONS: Pregnancy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- SV1, SV2 (Other): SV1 intervention: stroke volume using transthoracic echo SV2 intervention: stroke volume measured using the esCCO device.
  Interventions: Device: Transthoracic echo and esCCO stroke volume

INTERVENTIONS:
Device: Transthoracic echo and esCCO stroke volume — All participants will have their cardiac outputs measured using these two devices simultaneously. Cardiac output 1 will include measurements made using transthoracic echo and cardiac output 2 will be done using esCCO device.

SUMMARY:
Cardiac output (CO) is the volume of blood ejected from the heart and is a product of stroke volume (SV) vs heart rate (HR). It is closely related to Blood Pressure (BP) by the formula CO = Mean Arterial Pressure (MAP) / Systemic Vascular Resistance (SVR). Cardiac output monitoring is well established and validated for guiding fluid administration and resuscitation in intensive care and perioperatively in the non-pregnant population. Available CO monitoring methods may risk maternal health or fetal wellbeing or are unvalidated in the pregnant population. Invasive and semi-invasive methods of measuring CO such as the pulmonary artery catheter, the 'gold standard' require invasive arterial or central access negating their use in all but a select group of labouring women and have potentially serious risks attached to their usage. Echocardiography is a well-established and validated technique requiring no invasive access but the requirement for an experienced operator limits routine usage. It uses an external ultrasound probe to scan the heart.

Several novel non-invasive cardiac output monitors have recently come to the market including the estimated cardiac output esCCO monitor (Nihon Kohden) which uses Pulse Wave Transit Time (PWTT) to estimate cardiac output. It requires 3-lead Electrocardiography and pulse oximetry alone which is part of the routine monitoring for high risk patients on the labour ward.

The investigators research aims to evaluate the accuracy and precision of the esCCO in pregnant women and subsequently assess its utility during medical interventions such as epidural analgesia or caesarean section. The initial validation will take place in an antenatal clinic where women are assessed using Doppler echocardiography. The investigators will then compare the echocardiography results vs the esCCO results.

DETAILED DESCRIPTION:
The cardiac output (CO) is the volume of blood ejected by the heart each time it beats. It is the product of stroke volume (SV) and heart rate (HR) and is expressed in litres per minute. It gives a measure of the performance of the heart as a pump. The normal resting CO of a 70kg person is approximately 5 to 6 litres/min, due to a resting HR of 70-80 bpm multiplied by an average SV of 70-80ml. Different organs in the body receive differing proportions of the CO according to their demand. CO increases significantly in pregnancy due to the growing uterus, fetus and placenta, and its actual value can be affected by patient position and medical interventions, such as epidural analgesia.

Cardiovascular changes in pregnancy

During pregnancy, the cardiovascular system changes to adapt to the demands of the uteroplacental unit. CO starts to increase from the first trimester by 35-40%, to a 50% rise by the end of the second trimester. It remains at this level during the third trimester 1. The increase in CO occurs due to an increase in HR by up to 25% and SV by up to 30%. There is a further rise in CO during labour and delivery, which is transient.

CO also depends upon patient position, with a 13.5% increase in the left lateral position from supine. The increase in CO in the left lateral position is the basis for the left lateral tilt or wedge applied to the pregnant patient when supine. This reduces compression of the large abdominal blood vessels (aortocaval compression) by the gravid (pregnant) uterus and allows the CO to be maintained.

The proportion of the CO distributed to the uterus, kidneys and skin is greater in pregnancy compared to the non-pregnant state. Uterine blood flow is approximately 500 to 700 ml/min, which corresponds to 10-12% of the CO 1. More than 80% of this CO perfuses the placenta.

Lumbar epidurals in labour

Lumbar epidurals are used commonly for analgesia in labour, as well as for anaesthesia for operative interventions, such as lower segment Caesarean section (LSCS) and instrumental delivery. It is well known that epidural anaesthesia can cause haemodynamic changes, namely peripheral vasodilatation and a reduction in systemic vascular resistance (SVR) due to blockade of the sympathetic nervous system which controls many autonomic functions including blood pressure and heart rate 1. This can lead to a reduction in blood pressure if the CO is maintained, since the three are related by the formula; mean arterial pressure (MAP) = CO x SVR. If the CO drops, for example due to hypovolaemia (decreased amount of fluid in the circulation) or postural changes, then there will be a greater decrease in the blood pressure.

Valsalva manoeuvre Originally described in the 17th century, the Valsalva manoeuvre is performed by attempted exhalation against resistance, usually a closed airway. It is used routinely to equalize ambient pressure in the inner ear and sinuses ie during air travel or scuba diving. Medically it is used as a test of cardiac function and the autonomic nervous system which controls the hearts response to stimuli.

The standardised Valsalva manoeuvre requires a subject to be placed in a semirecumbent position and produce an expiratory pressure of 40mmHg for 10 seconds2.

Methods for measuring cardiac output There are several methods for measuring cardiac output, but their use in pregnancy may be limited by risks to mother or the effects of the technique on the developing fetus.

Invasive methods - The "gold standard" CO monitor is the pulmonary artery catheter. This measures CO using the temperature change of an injectate (the thermodilution principle) as blood is passing through the cardiac chambers. It is accurate and allows measurement of pulmonary artery pressures, but the obvious drawback is the invasive nature of the device, coupled with the risks of injury to the heart and pulmonary vessels. Due to its invasive nature, this is used almost exclusively in patients who are severely unwell, necessitating central catheterisation. Even so, there is currently no evidence from randomised controlled trials supporting the use of the pulmonary artery catheters 2. Its use is not possible in normal pregnancies, as it would be unacceptable to subject patients to the risks of central catheterisation. Other invasive techniques such as angiography or conductance catheters cause radiation exposure to the developing fetus.

Semi-invasive methods include LiDCO and PiCCO. The LiDCO monitor uses transpulmonary lithium dilution via a central line catheter and arterial sampling line for calibration. It then uses arterial waveform analysis to provide continuous CO measurements. PiCCO uses transpulmonary thermodilution, again via a central line and arterial sampling line. The disadvantages of these are that lithium dilution should be avoided in the first trimester and normal pregnancies do not require central or arterial lines. This negates their use in the normal pregnant population. However, newer LiDCO products such as the LiDCOrapid have been used in the literature 3.

Non-invasive methods for cardiac output measurement have been the cornerstone of studying maternal cardiac physiology in normal and pathological pregnancies in the last 20 years, since the introduction of Doppler echocardiography, around 1985 4. Echocardiographic techniques aim to estimate the SV, which can then be multiplied by the HR to obtain a CO value. This can be done using 2D, 3D or Doppler echocardiography 5. The obvious advantage is that no vascular access or calibration is needed, but an experienced operator is required, making routine use difficult.

Novel non-invasive cardiac output monitors have since appeared on the market, such as the noninvasive cardiac output monitor (NICOM), the ultrasonic cardiac output monitor (USCOM) and the estimated continuous cardiac output (esCCO) monitor.

The esCCO monitor The esCCO monitor is manufactured by Nihon Kohden6 and uses 3 lead electrocardiogram and a pulse oximeter (oxygen saturation probe) to estimate CO.

This method of measuring CO was shown to correlate well with the trend of CO measured using the pulmonary artery catheterisation method7, 8. It has also been shown to correlate well with the echo Doppler during exercise9. Bataille et al (2012) compared the esCCO monitor with transthoracic echocardiography for CO measurement in intensive care patients10. The authors deemed the esCCO to be clinically unacceptable in critically ill patients, although there were questions about the validity of this study11, 12. This is primarily because of extensive vasoconstriction and peripheral shut down with the critically ill septic patients. Use of this device in obstetrics is acceptable.

The esCCO monitor uses non-invasive blood pressure (NIBP), three-lead ECG and pulse oximetry (SpO2). These modalities are part of routine clinical monitoring, which makes this monitor ideal for measuring CO in the normal pregnant population. Patients admitted to the labour ward often require monitoring with at least NIBP and SpO2, hence only the three-lead ECG is 'extra'. By validating this monitor, CO measurement across a variety of clinical scenarios in the pregnant population will be possible.

ELIGIBILITY:
Inclusion Criteria:

* All consenting pregnant women above 18 years of age.

Exclusion Criteria:

* Women not consenting or unable to consent.
* Unwilling to remove nail varnish/false nails
* Peripheral circulatory problems eg Raynauds syndrome
* Unable to establish good plethysmography trace
* Medical conditions known to alter plethysmography eg hyperbiliruninaemia

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-11 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Comparison of stroke volume using esCCO monitor and trans thoracic echo in pregnant women | 30 minutes